CLINICAL TRIAL: NCT04152421
Title: Acceptability and Clinical, Cognitive and Brain Efficacy of the Pilot of a Computerized Psychotherapy Program Based on Behavioural and Cognitive Techniques in the Depressed Patient
Acronym: STOP DEPRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-AOI-05
Record Dates: First submitted 2019-10-24; First posted 2019-11-05 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Software user (Experimental)
  Interventions: Other: Software use

INTERVENTIONS:
Other: Software use — The patient will connect to a computerized platform to access the program. The program consists of 5 modules ("lessons"), each lasting approximately 40 minutes. Each module or lesson includes pedagogical assessments and explanations of the problem(s) in question, illustrations, testimonies, tips, exercises and recommended activities.

SUMMARY:
Depression is a common disease with a high rate of recurrence. It is a major public health problem with significant health costs. World Health Organization estimates that 34 million people worldwide are affected by depression but not treated. Common barriers to accessing care in depression would be: the high cost of therapy, long waiting times, low presence of therapists in some communities, travel difficulties, fear of being "stigmatized", not to mention the presence of negative biases towards psychotherapy. Behavioural and Cognitive Therapies are standardized psychotherapies using operationalized methodologies and offering a pedagogical approach to learning specific change techniques and skills. They are the treatment of choice for many of the mental disorders, including depression, which has been proven effective through numerous scientific studies. They are now recognized by the French Authority for Health as the most scientifically validated psychotherapies and are recommended in particular for the treatment of depression.

In a context of constant development of information technology and the Internet, computer programs and websites concerning health, and in particular mental health, have emerged. Among the mental health programs, Computer Based Cognitive Behavior Therapy programs in English-speaking countries now offer patients remote Internet-based behavioural and cognitive therapies.

These programs, which are not available in France, have been the subject of numerous meta-analyses demonstrating their therapeutic effectiveness. Some of these Computer Based Cognitive Behavior Therapy programs such as Beating The Blues® are recommended by health organizations such as the National Institute of Health and Clinical Excellence in the treatment of depression.

This advent of computerized therapies is part of a movement to raise awareness of the epidemiological extent of mood disorders and the inadequacy of management methods. These "therapist-free" programs are, via an interactive and multimedia interface, an alternative means of care, making it possible to overcome the usual obstacles to accessing care. In our opinion, they represent an important area of research in an increasingly computerized health system.

We propose to study the acceptability and effectiveness of the pilot of a Computer Based Cognitive Behavior Therapy targeting depression developed at the University of Nice Sophia Antipolis; in three dimensions:

1. Clinical: via scales for measuring depressive symptomatology and depression characteristics;
2. Cognitive: via specific scales of cognitive-behavioural dimensions and validated in depression.
3. Neurophysiological: via electroencephalographic markers linked to cognitive processes; The research framework would be that of a prospective trial. This work bridges the gap between neurosciences, neuropsychology and the psychiatric clinic, while at the same time being part of a commitment to research in the field of "e-health".

ELIGIBILITY:
Inclusion Criteria:

* French speaking
* Presenting a DSM 5 (Diagnostic and Statistical Manual of Mental Disorders, American Psychiatric Association) diagnosis of major depression
* Subject accepting the study and understanding its constraints

Exclusion Criteria:

* Patient at risk of suicide;
* Patient who does not meet the criteria for a major depressive episode;
* Patient meeting resistance depression criteria (Thase&Rush score > 3);
* Patient meeting the criteria for melancholic depression (DSM-5);
* Patient with "psychotic" elements within the depressive episode;
* Patient with chronic schizophrenic or psychotic comorbidity
* Patient with a depressive episode in bipolar disorder
* Patient with unbalanced epilepsy;
* Patient with a severe, unstable somatic condition;
* Patient with a cognitive impairment that hinders the proper use of the computer tool;
* Pregnant or birthing woman

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | 3 months
  The score varies from 0 to 39. 0 to 3: no depression 4 to 7: slight depression 8 to 15: medium to moderate depression 16 and over: severe depression

CONTACTS AND LOCATIONS:
Overall Officials: Bruno GIORDANA, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Hôpital Pasteur - Service de Psychiatrie, Nice, France